CLINICAL TRIAL: NCT05433987
Title: Study Aiming to Measure the Impact on Immune Activation and Inflammatory Markers of Switching From a Triple Combination Antiretroviral Therapy (cART) to a Long Acting Dual Therapy in HIV-infected Patients
Brief Title: Immune Activation Markers in HIV-infected Patients Switching to Long Acting Dual Therapy
Acronym: LONGADAPT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cannes Simone Veil (Other)
Responsible Party: Sponsor
Other Study IDs: CHC-PI-2022-01
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: HIV-1-infection
Keywords: inflammatory markers; dual therapy; treatment simplification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to measure the impact on immune activation and inflammatory markers of switching from a triple combination antiretroviral therapy (cART) to a long acting dual therapy in HIV-infected patients

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria will be offered to participate to the study.

In case of acceptance by given their writting consent, 6 ml of blood will be collected for measuring immune activation and inflammatory markers, during the blood test scheduled for the routine follow-up.

Six months after cART change, an equal volume of blood will be collected for measuring the same immune activation and inflammatory markers

ELIGIBILITY:
Inclusion Criteria:

* Patients agreeing to participate to the study and to collect their data
* HIV-1 infected subjects
* Patients switching from a stable (at least 6 months) and successful triple cART to a long acting dual cART
* Patients older than 18 yrs and regularly followed in Cannes and Nice hospitals
* Patients with a healthcare card

Exclusion Criteria:

* HIV-2 infected subjects
* Patients not being on successful and stable cART
* Patients having being treated during acute HIV-infection
* Patients modifying cART for virological failure
* Subjects modifying their treatment for another combination than from a triple cART to a dual cART
* Patients modifying cART during the 6 months of follow-up
* Patients refusing to participate to the study
* Patients included in an interventional study during the 6 months of follwo-up
* Patient under juridical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient HIV-1, regularly followed in Cannes and Nice Hospital and for which the doctor has decided to modify the treatment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Evolution the trajectory of immune activation and inflammatory markers | Baseline and 6 months after modiyfying cART
  Assess the trajectory of immune activation and inflammatory markers change at 6 month after modifying cART

SECONDARY OUTCOMES:
Prevalence of patients with successful cART | 1 month, 3 month, 6 month
  To evaluate prevalence of patients with successful cART (i.e. viral load below 50 copies/ml) 1 month after the switch

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Vassallo, MD, Principal Investigator — Centre Hospitalier de Cannes Simone Veil
Locations (1):
- Nathalie DOUX, Cannes, France